CLINICAL TRIAL: NCT04602429
Title: Children's Acute Surgical Abdomen Programme
Acronym: CASAP
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18/0342
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Children, Only; Surgery; Abdomen, Acute; Perioperative Complication
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the type and quality of care being delivered to children (aged 1 - 16 years old) undergoing emergency abdominal surgery in the United Kingdom by measuring baseline compliance against evidence-based recommendations and identifying variations in care between individual hospitals.

DETAILED DESCRIPTION:
The Children's Acute Surgical Abdomen Programme (CASAP) is a prospective national observational cohort study which aims to characterise the type and quality of care being delivered to children having emergency abdominal surgery.

The investigators aim to recruit every U.K. hospital undertaking this type of surgery in children, and capture information on 5000 patients over the study period.

The data collected will include information on patient risk factors, compliance with process quality indicators and the incidence and type of postoperative complications encountered. The data collected will be used to describe the current epidemiology of this patient group and to develop and internally validate a risk prediction tool for children undergoing emergency abdominal surgery. This tool be used to provide hospitals with their own risk-adjusted outcome measures and can subsequently be used to inform bedside decision-making. Patients will be followed up for 10 years through a data linkage process with National Health Service (NHS) Digital national databases.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 months and 16 years old
* Children undergoing unplanned abdominal surgery, where the preoperative diagnosis was considered to be related to a non-traumatic bowel (including appendix), hepatobiliary, and/or splenic pathology.

(Definitions - Unplanned is defined as non-elective (i.e. the patient presented requiring emergency or urgent intervention, either as a primary presentation or as a complication of previous surgery). Surgery is defined as a procedure undertaken by a surgeon in an operating theatre requiring the support of an anaesthetist. Any surgical approach (e.g. open, laparoscopic, robotic assisted etc) is acceptable.)

Exclusion Criteria:

* Patients / parents who do not provide consent.
* Children <12 months old on day of surgery
* Elective procedures
* Operations where the preoperative indication for surgery was considered to be traumatic, urological or gynaecological in origin
* Organ transplants
* Insertion/removal of dialysis catheters
* Interventional radiology procedures
* Caesarean sections
* Herniotomies, if the procedure does not involve access to the intra-abdominal cavity.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 - 16 years old undergoing emergency abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing postoperative morbidity. | 30 days
  Defined by the Clavien Dindo grading system:
  Grade I - Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Grade II - Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusions and total parenteral nutrition are also included. Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Intervention not under general anesthesia
  * IIIb Intervention under general anesthesia Grade IV Life-threatening complication (including Central Nervous System complications)* requiring Intensive Care Unit -management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgan dysfunction Grade V Death of a patient

SECONDARY OUTCOMES:
The length of hospital stay in days | 30 days
The number of patients who do not survive their in-hospital stay censored at 30 days. | 30 days
The mortality rate of children undergoing emergency abdominal surgery at 90 days, 1 year and 10 years post procedure date. | 90 days, 1 year and 10 years.
The readmission rate for children after having emergency abdominal surgery | 90 days and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Children's Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04602429/Prot_SAP_000.pdf